CLINICAL TRIAL: NCT03960606
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability, & Pharmacokinetics of Itraconazole Administered as a Dry Powder for Inhalation (PUR1900) in Asthmatic Patients With ABPA
Brief Title: Study in Adult Asthmatic Patients With Allergic Bronchopulmonary Aspergillosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 601-0014
Record Dates: First submitted 2019-05-14; First posted 2019-05-23 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary; Aspergillosis

STUDY DESIGN:
Intervention Model Description: Following screening and confirmation of eligibility, subjects will be randomly assigned (1:1:1:1) into 4 arms of 16 subjects each and will receive 10 mg, 20 mg, or 35 mg of PUR1900 or placebo, administered via dry powder inhalation daily for 28 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a double-blind manner. All study drug will be supplied in identical packaging and will be similar in color, smell, taste, and appearance to enable double-blind conditions. All study personnel will remain blinded until after database lock, unless the nature of their activities in the study specifically requires them to be unblinded. Any study documents, supplies, and tools will be reviewed to identify components that have the potential to unblind the study, and blinding restrictions will be applied where appropriate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 mg PUR1900 (Experimental): Study drug (PUR1900) will be administered orally, using a Dry Powder Inhaler (DPI) specific to the study (RS01 Monodose inhaler)
  Interventions: Combination Product: PUR1900
- 20 mg PUR1900 (Experimental): Study drug (PUR1900) will be administered orally, using a Dry Powder Inhaler (DPI) specific to the study (RS01 Monodose inhaler)
  Interventions: Combination Product: PUR1900
- 35 mg PUR1900 (Experimental): Study drug (PUR1900) will be administered orally, using a Dry Powder Inhaler (DPI) specific to the study (RS01 Monodose inhaler)
  Interventions: Combination Product: PUR1900
- Placebo (Placebo Comparator): Placebo
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: PUR1900 — PUR1900 contains itraconazole as the active ingredient, and it is formulated as a dry powder for oral inhalation.
  Arms: 10 mg PUR1900; 20 mg PUR1900; 35 mg PUR1900
Combination Product: Placebo — PUR1900 placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Multicenter, Placebo-Controlled, Phase 2 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Itraconazole Administered as a Dry Powder for Inhalation (PUR1900) in Adult Asthmatic Patients With Allergic Bronchopulmonary Aspergillosis

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, placebo controlled, multiple-arm study.

Following screening and confirmation of eligibility, subjects will be randomly assigned (1:1:1:1) into 4 arms of 16 subjects each and will receive 10 mg, 20 mg, or 35 mg of PUR1900 or placebo, administered via dry powder inhalation daily for 28 days. The doses of PUR1900 are stated in this protocol as the respective nominal doses of itraconazole.

Subject eligibility for the study will be determined within 28 days before the first dose of study drug (Day 1) and will be confirmed between 9 and 6 days before dosing and again on Day 1.

Eligible subjects will begin daily dosing with study drug (PUR1900 or placebo) on Day 1.

Subjects will return to the study site for visits on Days 2, 7, 14, and 28 and will be dosed at the study site. The remaining daily doses of study drug will be self-administered at home.

A follow-up visit will occur 7 to 10 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female, 18 to 75 years old (inclusive) at the time of signing the informed consent.
* Has a body mass index of 18.0 to 35.0 kg/m2 (inclusive) at screening.
* Has a historical diagnosis of asthma, as per the Global Initiative for Asthma (GINA) 2018 update.
* Has a confirmed historical diagnosis of ABPA, as per the Modified International Society for Human and Animal Mycology (ISHAM) working group 2013 criteria.
* Is currently considered to be in one of the following stages of ABPA: Stage 2 (Response), Stage 4 (Remission), Stage 5a (Treatment-dependent ABPA), or Stage 5b (Glucocorticoid-dependent asthma)
* Has a serum immunoglobulin (Ig) E ≥1000 IU/mL during screening (Visit 1 or Visit 2).
* Can perform a valid, reproducible spirometry test with demonstration of a prebronchodilator FEV1 ≥50% of predicted normal for age, sex, race, and height (Quanjer et al 2012) at a screening visit.
* Has a documented stable asthma medication regimen during screening (Day 28 to Day 1), including SABA, LABA, and LTRA use and inhaled and/or oral GCS.
* Subjects who are sexually active, male subjects able to father a child, and female subjects of childbearing potential must agree to follow the contraception requirements of this protocol.
* Can demonstrate the correct inhalation technique for the use of the delivery device at screening and before dosing.

Exclusion Criteria:

* Is a female of childbearing potential who is pregnant or lactating or who plans to become pregnant during the study. A woman is considered to be of childbearing potential unless she is either permanently sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion/ligation) or postmenopausal (had no menses for 12 months without an alternative medical cause).
* Has a history of life-threatening asthma within the last 5 years, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, and/or hypoxic seizures.
* Had an occurrence of asthma or ABPA exacerbations within the 28 days before screening or during the 28-day period before Day 1.
* Had an occurrence of clinically significant bacterial, viral, or fungal infection that required systemic (oral or intravenous) antibiotics, antivirals, or antifungals within the 28 days before screening. Topical treatments, other than antifungals, are allowed.
* Received any investigational medical product in a clinical research study within the previous 3 months before dosing in this study.
* Has previously received PUR1900.
* Has a history of any significant drug or alcohol abuse in the past 2 years before screening, as judged by the investigator.
* Has current tobacco or inhaled marijuana use or history of smoking tobacco or marijuana within the last 6 months before screening.
* Is a current user of e-cigarettes or has used these products within the last 6 months before screening.
* Has a positive urine test result for drugs of abuse, alcohol, or cotinine at screening
* Has a history of allergies to or hypersensitivity reactions after dosing of itraconazole or other antifungal azoles.
* Had a major trauma or surgery within the last 28 days before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
Incidence of intraday FEV1 declines | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
Respiratory rate | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
Blood pressure | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  Systolic pressure over diastolic pressure
Heart rate | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  Beats per minute
Oxygen saturation | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  As a percentage
Physical examination findings | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  Physician's notes
Clinical laboratory test results | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  Lab reports with any out of range results flagged
12-Lead electrocardiogram findings | From Day 1 through Follow Up (which is 7 to 10 days after the last dose)
  ECG report and tracing

SECONDARY OUTCOMES:
Sputum concentrations of itraconazole and hydroxy-itraconazole | Day 2 to Day 28
Sputum eosinophils | (Day -9 to Day -6) to Day 28
To evaluate the effect of PUR1900 on pulmonary function following single- and multiple-dose administration of PUR1900 | Day 1 to Day 28
Asthma Control Questionnaire-6 (ACQ 6) | Day 1 to Day 28
  Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
Change from baseline (Day 1) to Day 28 in A fumigatus burden in sputum | Day 1 to Day 28
  As assessed by quantitative PCR and sputum culture
Cmax (maximum observed concentration in plasma) | Day 1 to Day 28
Tmax (time to maximum concentration in plasma) | Day 1 to Day 28
AUC (area under the concentration-time curve) | Day 1 to Day 28
CL/F (clearance) | Day 1 to Day 28
Vz/F (apparent volume of distribution) | Day 1 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: William J. Calhoun, MD, Principal Investigator — University of Texas Medical Branch Galveston, TX 77555; David Denning, FRCP, FRC Path, FIDSA, FMedSci, Principal Investigator — Director, National Aspergillosis Centre Manchester, Wythenshawe M23 9LT, UK
Locations (20):
- United States (9):
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Integrity Clinical Research Center Inc., Hialeah, Florida
  - Heuer M.D Research Inc., Miami Lakes, Florida
  - Infinite Clinical Trials, Roswell, Georgia
  - University Consultants In Allergy and Immunology, Chicago, Illinois
  - Laporte County Institute for Clinical Research, Michigan City, Indiana
  - Montefiore Medical Center, The Bronx, New York
  - University of Texas Medical Branch at Galveston, Galveston, Texas
- Australia (2):
  - John Hunter Hospital, New Lambton, New South Wales
  - Mater Private Hospital Brisbane, Brisbane, Queensland
- India (3):
  - Yashoda Hospital, Hyderabad, Andhra Pradesh
  - Shree Hospital And Critical Care Centre, Nagpur, Maharashtra
  - SMS Medical College and Hospital, Jaipur, Rajasthan
- Poland (4):
  - Centrum Alergologii Teresa Hofman, Poznan, Greater Poland Voivodeship
  - Centrum Medycyny Oddechowej Mroz sp. j., Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne - PPDS, Gdansk, Pomeranian Voivodeship
  - PULMAG Arkadiusz Brodowski, Grzegorz Gasior S. C., Sosnowiec, Silesian Voivodeship
- United Kingdom (2):
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Wythenshawe Hospital - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: No